CLINICAL TRIAL: NCT06744374
Title: An Observational, Non-Interventional Comparative Effectiveness Study of Mortality Outcomes and Related Cardiopulmonary Events Among a Cohort of Commercially Insured Chronic Obstructive Pulmonary Disease (COPD) Patients Who Initiate Breztri and Multiple Inhaler Triple Therapy (MITT) in the United States (US)
Brief Title: A Comparative Effectiveness Study of Mortality Outcomes and Related Cardiopulmonary Events Among a Cohort of Chronic Obstructive Pulmonary Disease (COPD) Patients Who Initiate Breztri and Multiple Inhaler Triple Therapy (MITT) in the United States (US)
Acronym: SKOPOS:MAZI
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D5980R00098
Record Dates: First submitted 2024-12-17; First posted 2024-12-20 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Pulmonary Disease, Chronic Obstructive
Keywords: COPD; Retrospective; Observational; Triple Therapy; Cardiopulmonary; Mortality
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- COPD Patients: COPD patients initiating BGF or MITT
  Interventions: Drug: BGF; Drug: MITT

INTERVENTIONS:
Drug: BGF — Budesonide/glycopyrrolate/formoterol fumarate
  Other Names: Breztri
Drug: MITT — Multiple-inhaler triple therapy
  Other Names: Open triple therapy combination

SUMMARY:
Patients with chronic obstructive pulmonary disease (COPD) have elevated risk of mortality and cardiopulmonary events, particularly following exacerbations. While single inhaler triple therapies (SITTs), such as budesonide/glycopyrrolate/formoterol fumarate (BGF), reduce mortality and cardiopulmonary event risk versus dual bronchodilator therapy, there is limited evidence comparing outcomes associated with SITTs versus multiple inhaler triple therapies (MITTs). SKOPOS-MAZI was a retrospective comparative effectiveness study in patients with COPD aged ≥40 years using US administrative claims data from Optum's de-identified Clinformatics® Data Mart Database. The primary and secondary endpoints were time to all-cause mortality (ACM) and time to first severe cardiopulmonary event following initiation of BGF or MITT (identification period: October 1, 2020-June 30, 2023; index date: first prescription fill). Relative hazards of outcomes were assessed until a censoring event using Cox proportional hazards models, with inverse propensity treatment weighting accounting for between-group imbalances (standardized mean difference >0.1) in baseline characteristics.

ELIGIBILITY:
Inclusion Criteria:

* 1 initial prescription for BGF or MITT starting October 1, 2020 through to the latest available data update, AND

  * Age ≥40 years on date of first prescription for BGF or MITT episode, AND
  * Continuous medical and pharmacy health plan eligibility for ≥12-months (365 days) prior to first prescription for BGF or MITT AND
* 2 medical claims with diagnoses for COPD at least 30 days apart occurring on or anytime in the patient's available 24-month history before the first BGF prescription or MITT episode, with one diagnosis occurring in the immediate 12-month period prior to or on initiation of BGF or MITT

Exclusion Criteria:

* Age <40 at time of treatment initiation
* Invalid or unknown gender
* If death date occurs prior to or on study index date
* <12 months (365 days) of medical and pharmacy health plan eligibility/coverage prior treatment initiation
* Presence of ≥1 prescription claim for any triple therapy during the patient's entire available baseline history (BGF, FF/UMEC/VI or MITT)
* "potential MITT use" in baseline, MITT for baseline purposes will be defined as ≥1 days continuous days where all three MITT components (ICS, LABA, LAMA) are observed in combination (dual + monotherapy) or as three separate monotherapy components
* History of any of the following conditions, procedures or events during the immediate baseline 12-month period: (a) ≥1 medical claim (i.e., office, ED or hospital) in any position with a diagnosis for alpha-1-antitrypsin deficiency, interstitial fibrosis, lung cancer, pulmonary embolism, sarcoidosis; (b) ≥1 medical claim for hospice services; (c) Any medical Bill Type Code (BILL_TYPE_CODE ) starting with 81 or 82; or Revenue codes (RVNU_CD): 0651-0659; (d) ≥1 medical claim with a diagnosis code of encounter related to clinical trial participation (Z00.6) at any point during the study period (including both baseline and follow-up periods)

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Commercially insured (including Medicare Advantage) patients diagnosed with COPD captured in the Optum CDM who are ≥40 years of age at the time of triple therapy initiation and who have at least two medical claim diagnoses for COPD (J41-J44) occurring on two separate occasions ≥30 days apart. Patients included will be new initiators of triple therapy (BGF or MITT) and have no record of a prescription fill for any triple therapy (including FF/UMEC/VI) during their entire available baseline history with at least the 12 months baseline history available prior to their first observed prescription for BGF or MITT
Sampling Method: Non-Probability Sample
Enrollment: 22369 (Actual)
Dates: Start 2024-02-29 (Actual); Primary Completion 2024-03-30 (Actual); Study Completion 2024-03-30 (Actual)

PRIMARY OUTCOMES:
Time to and rate of all-cause mortality | During available follow-up; median 313 days
  Time to and rate of all-cause mortality observed after initiation of BGF or MITT; all-cause mortality as defined by the available death information contained in the database.

SECONDARY OUTCOMES:
Time to and rate of cardiopulmonary events | During available follow-up; median 313 days
  Time to and rate of cardiopulmonary events observed during the follow-up period after initiation of BGF or MITT; cardiopulmonary events defined as a composite measure of severe (hospitalizations) COPD exacerbations and MACE-related events, and all-cause mortality

CONTACTS AND LOCATIONS:
Overall Officials: Michael Pollack, MS, Study Chair — AstraZeneca
Locations (1):
- AstraZeneca, Wilmington, Delaware, United States

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal Vivli.org. All requests will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
  Yes, indicates that AZ are accepting requests for IPD, but this does not mean all requests will be shared.
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA PhRMA Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the anonymized individual patient-level data via secure research environment Vivli.org. Signed Data Usage Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information.
URL: https://vivli.org/

REFERENCES:
- See also: D5980R00098_CSR synopsis_Redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D5980R00098&attachmentIdentifier=76f19dd8-1b0f-4688-9014-30bafe9b9f93&fileName=D5980R00098_Clinical_Study_Report_synopsis_Redacted.pdf&versionIdentifier=